CLINICAL TRIAL: NCT02454361
Title: A Randomized, Double-blind, Placebo-controlled, Sequential Parallel Group, Single Ascending Dose Study in Healthy Subjects to Evaluate the Safety, Tolerability and Pharmacokinetics of KBP-7072 Following Oral Administration
Brief Title: Safety, Tolerability and Pharmacokinetics of KBP-7072
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KBP Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KBP7072-1-001
Record Dates: First submitted 2015-05-18; First posted 2015-05-27 (Estimated); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: Safety; tolerability; pharmacokinetics; KBP-7072
MeSH Terms: interventions — kbp-7072

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- KBP-7072 cohort 1 (Experimental): KBP-7072 by mouth once
  Interventions: Drug: KBP-7072; Drug: Placebo
- KBP-7072 cohort 2 (Experimental): KBP-7072 by mouth once
  Interventions: Drug: KBP-7072; Drug: Placebo
- KBP-7072 cohort 3 (Experimental): KBP-7072 by mouth once
  Interventions: Drug: KBP-7072; Drug: Placebo
- KBP-7072 cohort 4 (Experimental): KBP-7072 by mouth once
  Interventions: Drug: KBP-7072; Drug: Placebo
- KBP-7072 cohort 5 (Experimental): KBP-7072 by mouth once
  Interventions: Drug: KBP-7072; Drug: Placebo
- KBP-7072 Fed Group (Experimental): KBP-7072 by mouth once to the fed group
  Interventions: Drug: KBP-7072

INTERVENTIONS:
Drug: KBP-7072 — KBP-7072
Drug: Placebo — Placebo
  Arms: KBP-7072 cohort 1; KBP-7072 cohort 2; KBP-7072 cohort 3; KBP-7072 cohort 4; KBP-7072 cohort 5

SUMMARY:
This is a randomized, double-blind, placebo-controlled, dose-escalation study to evaluate the safety, tolerability and pharmacokinetics of a single dose of KBP-7072 following oral single ascending dose administration and with an open label food effect panel.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, dose-escalation study to evaluate the safety, tolerability and pharmacokinetics of a single dose of KBP-7072 following oral single ascending dose administration and with an open label food effect panel.

Part 1: A total of 40 subjects will be evaluated with 30 subjects randomized to receive active drug and 10 subjects randomized to receive placebo in a double-blind fashion (eight subjects in each dose cohort, six subjects randomized to active drug and two subjects randomized to placebo). 5 dose levels will be evaluated. Extensive PK samplings will be collected after dosing (pre-dose (within 30 min prior to dosing) and at 0.5, 1, 2, 4, 6, 10, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216 and 240 hr post-dose).

Part 2: A separate panel of 6 subjects will receive a single dose of KBP-7072 under fed conditions. The dose tested in Part 2 will be determined based on the safety, tolerability and PK data available from Part 1. Extensive PK samplings will be collected after dosing (pre-dose (within 45 min prior to dosing) and at 0.5, 1, 2, 4, 6, 10, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216 and 240 hr post-dose).

Safety assessments will include monitoring of adverse events (AEs), vital signs (blood pressure, pulse rate, respiratory rate and oral temperature), clinical laboratory findings, 12-lead electrocardiograms (ECGs), and physical examination findings.

ELIGIBILITY:
Inclusion Criteria:

* males and surgically sterile or postmenopausal females
* aged between 18-45 years
* body mass index (BMI) 19 ≤ BMI ≤ 30 kg/m2,
* no significant medical history
* normal renal function
* good general health

Exclusion Criteria:

* Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, pulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability (i.e., number of participants with adverse events): predose and postdose | 10 days

SECONDARY OUTCOMES:
Area Under Curve (AUC) Time Frame: predose, 0.5, 1, 2, 4, 6, 10, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216 and 240 hr post-dose | 10 days
Area Under Curve (AUC) Time Frame: predose, 0.5, 1, 2, 4, 6, 10, 12, 18, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216 and 240 hr post-dose among participants who have had food | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- KBP, Princeton, New Jersey, United States

REFERENCES:
- [Derived] Huband MD, Mendes RE, Pfaller MA, Lindley JM, Strand GJ, Benn VJ, Zhang J, Li L, Zhang M, Tan X, Liu Q, Flamm RK. In Vitro Activity of KBP-7072, a Novel Third-Generation Tetracycline, against 531 Recent Geographically Diverse and Molecularly Characterized Acinetobacter baumannii Species Complex Isolates. Antimicrob Agents Chemother. 2020 Apr 21;64(5):e02375-19. doi: 10.1128/AAC.02375-19. Print 2020 Apr 21. PMID 32071042